CLINICAL TRIAL: NCT00775190
Title: Side Effect Profiles of Brand Name Versus Generic Oral Contraceptives
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unale to recruit , progress report not filed by PI
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, John Uckele, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2008-184
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Contraception
Keywords: birth control pills; oral contraceptives; brand name; generic; side effects; oral contraceptive side effects; dysfunctional uterine bleeding; pre-menstrual symptoms
MeSH Terms: conditions — Metrorrhagia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ortho tricyclen™ (Active Comparator): Participant Randomized to Ortho tricyclen 1 tablet by mouth Daily
  Interventions: Drug: ortho tricyclen
- Trinessa™ (Active Comparator): Participant Randomized to Trinessa 1 tablet by mouth Daily
  Interventions: Drug: Trinessa

INTERVENTIONS:
Drug: ortho tricyclen — brand name oral contraceptive
  Arms: Ortho tricyclen™
Drug: Trinessa — generic oral contraceptive
  Arms: Trinessa™

SUMMARY:
This is a randomized control trial of Ortho tricyclen versus Trinessa (generic equivalent) to determine if they have similar effects. Women will be randomized to receive either Ortho tricyclen or Trinessa oral contraceptives and will be asked to keep a daily dairy of any symptoms or bleeding experienced. Once a month, participants will be asked to complete a survey.

The objective is to compare generic oral contraceptives (OCPs) and brand name OCPs with respect to side effect profiles including bleeding patterns, mood changes, nausea and vomiting, frequency of menstrual cramps, breast tenderness, elevation in blood pressure, stroke, blood clots and patient compliance.

DETAILED DESCRIPTION:
This is a double blind randomized controlled trial of Ortho tricyclen™ vs. Trinessa™ (generic equivalent) to determine if they have similar effects on bleeding patterns, namely days of menstrual flow, amount of bleeding, and intermenstrual bleeding. Women will score these parameters using a survey with objective measures for days of bleeding, amount of flow, and days of breakthrough bleeding. As secondary outcomes, we will compare the side effect profiles of each in regards to nausea, vomiting, breast tenderness, menstrual cramps, mood changes, and thromboembolic events.

Patients will record in their daily diary if one of the outcomes occurs or not. We will observe whether the events occur and the number of occurrences within the six month time period.

ELIGIBILITY:
Inclusion Criteria:

* nonsmoker
* not pregnant
* not planning to become pregnant in the next 6 months
* not taking hormonal birth control for at least 3 months previous to entering the study
* no history of fibroids
* no history of ovarian cysts
* no history of dysfunctional uterine bleeding

Exclusion Criteria:

* pregnant
* under the age of 18
* over the age of 35
* history of irregular uterine bleeding
* history of ovarian cysts
* history of fibroids
* history of migraines with aura
* history of liver disease
* family or personal history of Blood clots (thromboembolism)
* mental disabilities
* desire to become pregnant in the next six months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Bechek, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ortho Tricyclen™ | Trinessa™
Started | 7 | 5
Completed | 3 | 0
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ortho Tricyclen™ | Trinessa™ | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] — target population females ages 18-65
  years | 24 [21 to 31] | 24 [21 to 31] | 24 [21 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Beaumont Health System patient population
  participants
    United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Amount of Bleeding
Description: Measures how light or heavy the menstrual flow on a 1 to 3 Likert scale. (Light, Medium, Heavy).
Time Frame: 6 Months
Population: Study Terminated with no data analysis.
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Incidence of Breakthrough Bleeding
Description: Any breakthrough bleeding during reporting period.
Time Frame: 6 months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Days of Bleeding
Description: Number of days with bleeding during each menstrual period.
Time Frame: 6 months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Side Effects (Nausea)
Description: Number of days of nausea
Time Frame: 6 months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Side Effects (Vomiting)
Description: Number of episodes of vomitting
Time Frame: 6 Months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Side Effects (Breast Tenderness)
Description: Incidence of breast tenderness during the study time frame
Time Frame: 6 Months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Side Effects (Mood Changes)
Description: Self reported changes in mood during each month over the time frame.
Time Frame: 6 months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Side Effects (Menstrual Cramps)
Description: Intensity of menstrual cramps reported on a 4 point Likert scale.
Time Frame: 6 months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Side Effects (Incidence of Thromboembolic Events)
Description: Occurrence of any thromboembolic events during the study time frame.
Time Frame: 6 months
Population: Study Terminated with no data analysis
Arm/Group | Ortho Tricyclen™ | Trinessa™
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ortho Tricyclen™ | Trinessa™
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

LIMITATIONS AND CAVEATS:
Early Study termination. No data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes